CLINICAL TRIAL: NCT07313956
Title: Mode of Ventilation During Critical Illness at Multiple Centers
Acronym: MODEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin P Seitz, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 250596; K23HL175246 (NIH)
Record Dates: First submitted 2025-12-30; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Failure; Mechanical Ventilation; Critical Illness
MeSH Terms: conditions — Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Intervention Model Description: In the MODEM trial, the entire study ICU will be assigned to a single ventilator mode (cluster-randomized) and the ICU will switch between volume control, pressure control, and adaptive pressure control modes every two months in a randomly generated sequence (cluster-crossover). Enrolled patients will be assigned to only one group at the time of their enrollment.
Masking Description: Observer bias will be minimized by use of objective endpoints collected in duplicate by [1] study personnel and [2] automated data extraction from the electronic health record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adaptive Pressure Control Group (Active Comparator): During invasive mechanical ventilation in a study location, adaptive pressure control will be used as the mode for continuous mandatory ventilation.
  Interventions: Other: Adaptive pressure control
- Pressure Control Group (Active Comparator): During invasive mechanical ventilation in a study location, pressure control will be used as the mode for continuous mandatory ventilation.
  Interventions: Other: Pressure control
- Volume Control Group (Active Comparator): During invasive mechanical ventilation in a study location, volume control will be used as the mode for continuous mandatory ventilation.
  Interventions: Other: Volume control

INTERVENTIONS:
Other: Volume control — Volume control mode for invasive mechanical ventilation
  Arms: Volume Control Group
Other: Pressure control — Pressure control mode for invasive mechanical ventilation
  Arms: Pressure Control Group
Other: Adaptive pressure control — Adaptive pressure control for invasive mechanical ventilation
  Arms: Adaptive Pressure Control Group

SUMMARY:
The goal of this clinical trial is to learn whether the choice of ventilator mode for patients on breathing machines in the intensive care unit affects their survival and recovery. To do this, researchers will assign the entire participating intensive care unit to one of the three available ventilator modes, alternating which mode is assigned in random sequence every 2 months. The main question it aims to answer is: Does the choice between volume control, pressure control, and adaptive pressure control affect the number of days that patients are alive and free of the breathing machine?

DETAILED DESCRIPTION:
The MODEM trial is a cluster-randomized, cluster-crossover clinical trial comparing the effectiveness of three ventilator modes (volume control vs pressure control vs adaptive pressure control) for mechanical ventilation of critically ill adults at multiple centers. A total of 4,785 critically ill adults receiving invasive mechanical ventilation in intensive care units will be enrolled and included in the primary analysis. Each study unit will be assigned to a ventilator mode and will switch between modes every 2 months in an order determined by randomization. Enrolled patients will be assigned to receive volume control, pressure control, or adaptive pressure control according to the mode assigned to the unit at the time they were enrolled. The primary outcome will be ventilator-free days in the first 28 days, and the secondary outcome will be all-cause, 28-day in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient is receiving mechanical ventilation through an endotracheal tube or tracheostomy
* Patient is physically located in a participating adult ICU

Exclusion Criteria:

* Patient is known to be less than 18 years old
* Patient is known to be a prisoner
* Patient is known to have been receiving invasive mechanical ventilation at place of residence prior to hospital admission
* Patient is receiving extracorporeal membrane oxygenation at the time when inclusion criteria are first met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4785 (Estimated)
Dates: Start 2027-07 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days in the first 28 days | From enrollment to 28 days after enrollment
  The number of calendar days between enrollment and 28 days after enrollment, on which the patient is alive and free of invasive mechanical ventilation. Receipt of invasive mechanical ventilation will be considered to end when patients undergo the final tracheal extubation or disconnection of the ventilator from a tracheostomy tube between enrollment and day 28.

SECONDARY OUTCOMES:
All-cause, 28-day, in-hospital mortality | From enrollment to 28 days after enrollment
  All-cause, 28-day, in-hospital mortality, defined as death from any cause occurring between enrollment and 28 days after enrollment with outcome ascertainment ending at hospital discharge.

OTHER OUTCOMES:
Severe acidemia (Safety Outcome) | From enrollment to 28 days after enrollment
  pH <7.1 on blood gas laboratory test
Barotrauma (Safety Outcome) | From enrollment to 28 days after enrollment
  Pneumothorax or pneumomediastinum
Receipt of invasive procedure for treatment of pneumothorax or pneumomediastinum (Safety Outcome) | From enrollment to 28 days after enrollment
  E.g., thoracostomy tube
Shock (Safety Outcome) | From enrollment to 28 days after enrollment
  Receipt of continuous infusion of vasopressor or inotrope medications
Exhaled tidal volume (Exploratory Intermediary Outcome) | From enrollment to 28 days after enrollment
  Measured in mL/kg of predicted body weight
Exhaled tidal volumes above target range (Exploratory Intermediary Outcome) | From enrollment to 28 days after enrollment
  Proportion of recorded breaths with exhaled tidal volume values above the target range (>8 mL/kg predicted body weight)
Peak inspiratory pressure (Exploratory Intermediary Outcome) | From enrollment to 28 days after enrollment
  Measured in cmH2O
Peak inspiratory pressures above target range (Exploratory Intermediary Outcome) | From enrollment to 28 days after enrollment
  Proportion of recorded breaths with peak inspiratory values above the target range (>30cmH2O)
Richmond Agitation-Sedation Scale (RASS) (Exploratory Intermediary Outcome) | From enrollment to 28 days after enrollment
Deep sedation (Exploratory Intermediary Outcome) | From enrollment to 28 days after enrollment
  Proportion of assessments with RASS of -4 or -5
Delirium and coma-free days in the first 28 days (Exploratory Clinical Outcome) | From enrollment to 28 days after enrollment
  The number of calendar days between enrollment and 28 days after enrollment, on which the patient is alive and free of delirium or coma
Intensive care unit-free days in the first 28 days (Exploratory Clinical Outcome) | From enrollment to 28 days after enrollment
  The number of calendar days between enrollment and 28 days after enrollment, on which the patient is alive and free from intensive care unit admission after the final transfer out of the intensive care unit
Hospital free days in the first 28 days (Exploratory Clinical Outcome) | From enrollment to 28 days after enrollment
  The number of calendar days, between enrollment and 28 days after enrollment, on which the patient is alive and free from hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Rappaport SH, Shpiner R, Yoshihara G, Wright J, Chang P, Abraham E. Randomized, prospective trial of pressure-limited versus volume-controlled ventilation in severe respiratory failure. Crit Care Med. 1994 Jan;22(1):22-32. doi: 10.1097/00003246-199401000-00009. PMID 8124968
- [Background] Esteban A, Alia I, Gordo F, de Pablo R, Suarez J, Gonzalez G, Blanco J. Prospective randomized trial comparing pressure-controlled ventilation and volume-controlled ventilation in ARDS. For the Spanish Lung Failure Collaborative Group. Chest. 2000 Jun;117(6):1690-6. doi: 10.1378/chest.117.6.1690. PMID 10858404
- [Background] Rittayamai N, Katsios CM, Beloncle F, Friedrich JO, Mancebo J, Brochard L. Pressure-Controlled vs Volume-Controlled Ventilation in Acute Respiratory Failure: A Physiology-Based Narrative and Systematic Review. Chest. 2015 Aug;148(2):340-355. doi: 10.1378/chest.14-3169. PMID 25927671
- [Background] Chatburn RL, El-Khatib M, Mireles-Cabodevila E. A taxonomy for mechanical ventilation: 10 fundamental maxims. Respir Care. 2014 Nov;59(11):1747-63. doi: 10.4187/respcare.03057. Epub 2014 Aug 12. PMID 25118309
- [Background] Telias I, Madorno M, Pham T, Coudroy R, Mellado Artigas R, Baedorf-Kassis E, Chen CW, Spadaro S, Chiumello D, Beitler J, Kondili E, Tiribelli N, Fredes S, Becher T, Dres M, Liu K, Terzi N, Guerin C, Mauri T, Roca O, Mancebo J, Rodriguez N, Arnal JM, Goligher EC, Diehl JL, Jochmans S, Beloncle F, Rittayamai N, Mojoli F, Heunks L, de Vries H, Zhou JX, Guervilly C, Brochard L. Physiological Consequences of Breathing Effort According to the Mode of Ventilation During Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2025 Jul 23. doi: 10.1164/rccm.202411-2155OC. Online ahead of print. PMID 40700741
- [Background] Seitz KP, Lloyd BD, Wang L, Shotwell MS, Qian ET, Muhs AL, Richardson RK, Rooks JC, Hennings-Williams V, Sandoval CE, Richardson WD, Morgan TL, Thompson AN, Hastings PG, Ring TP, Stollings JL, Talbot EM, Krasinski DJ, DeCoursey BR, Marvi TK, DeMasi SC, Gibbs KW, Self WH, Mixon AS, Rice TW, Semler MW, Casey JD; Pragmatic Critical Care Research Group. Effect of Ventilator Mode on Ventilator-Free Days in Critically Ill Adults: A Randomized Clinical Trial. Chest. 2025 Oct;168(4):912-923. doi: 10.1016/j.chest.2025.03.024. Epub 2025 Apr 4. PMID 40189043